CLINICAL TRIAL: NCT02564497
Title: A Randomized, Open-label, Parallel-group, Single-dose, Biocomparability Study of the Pharmacokinetics of Belatacept Drug Products Using Active Pharmaceutical Ingredient Manufactured by Process E Relative to Active Pharmaceutical Ingredient Manufactured by Process C in Healthy Subjects
Brief Title: A Study to Compare the Pharmacokinetics of Belatacept Using Active Pharmaceutical Ingredient Manufactured by Process E Relative to Process C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IM103-349
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-12

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Process E Belatacept (Other): Active Pharmaceutical Ingredient (API) of Belatacept manufactured by Process E
  Interventions: Biological: Process E Belatacept
- Process C Belatacept (Other): Active Pharmaceutical Ingredient (API) of Belatacept manufactured by Process C
  Interventions: Biological: Process C Belatacept

INTERVENTIONS:
Biological: Process E Belatacept
  Arms: Process E Belatacept
Biological: Process C Belatacept
  Arms: Process C Belatacept

SUMMARY:
The purpose of the study is to compare the Pharmacokinetics (PK) of Process E belatacept relative to Process C belatacept in Healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy males and females.
3. Males and females, ages 18 to 55 years, inclusive.
4. Women of child bearing potential (WOCBP) with negative serum or urine pregnancy test
5. Women must not be breastfeeding
6. Men and WOCBP must agree to follow instructions for contraception

Exclusion Criteria:

1. History of TB, malignancy, any other chronic or acute infecton or disease.
2. History of acute or chronic medical illness
3. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population.
4. History of allergy to belatacept or related compounds -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 491 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2017-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 491 participants were enrolled; 146 were randomized and treated. 232 participants were enrolled but not randomized because they no longer met study criteria, 1 participant withdrew consent and 112 participants were not randomized for other reasons.
Period: Overall Study
Arm/Group | Process E Belatacept | Process C Belatacept
Started | 74 | 72
Completed | 74 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Process E Belatacept | Process C Belatacept | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.60) | 35.4 (10.48) | 34.5 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 68
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 42 | 91
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    Overall Participants: White | 58 | 56 | 114
    Overall Participants: Black or African American | 14 | 14 | 28
    Overall Participants: American Indian or Alaskan Native | 1 | 0 | 1
    Overall Participants: Asian | 0 | 1 | 1
    Overall Participants: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Overall Participants: Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero Extrapolated to Infinite Time (INF) of Belatacept.
Description: (AUC[INF]) was derived from serum concentration versus time data and measured in nanogram hours per milliliter (ng*h/mL). Serum samples were analyzed for belatacept by a validated enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
ng.h/mL | 17084539 (17) | 21579398 (17)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Belatacept
Description: Cmax was derived from serum concentration versus time data. Serum samples were analyzed for belatacept by a validated enzyme-linked immunosorbent assay (ELISA). Cmax was measured in nanograms per milliliter.
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
ng/mL | 269305 (16) | 255169 (16)

3. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Tmax was derived from serum concentration versus time data. Serum samples were analyzed for belatacept by a validated enzyme-linked immunosorbent assay (ELISA). Tmax was measured in hours (h).
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Median (90% Confidence Interval); unit: h
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
h | 1.00 [0.467 to 2.00] | 1.00 [0.467 to 2.00]

4. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC 0-T)
Description: (AUC[0-T]) was derived from serum concentration versus time data and measured in nanogram hours per milliliter (ng.h/mL). Serum samples were analyzed for belatacept by a validated enzyme-linked immunosorbent assay (ELISA)
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
ng.h/mL | 17020284 (16) | 21422168 (16)

5. Secondary Outcome: Total Body Clearance (CLT)
Description: CLT was the volume of belatacept cleared by the system, normalized by baseline body weight. Serum samples were analyzed for belatacept by a validated enzyme-linked immunosorbent assay (ELISA). CLT was measured in liters per hour.
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
L/h | 0.0433 (18) | 0.0343 (19)

6. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
L | 7.89 (15) | 7.35 (19)

7. Secondary Outcome: Half Life (T-HALF)
Time Frame: Day 1 to Day 71
Population: All randomized, treated participants with evaluable PK data
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Process E Belatacept | Process C Belatacept
Number analyzed (Participants) | 73 | 72
h | 160 (39.5) | 183 (47.7)

ADVERSE EVENTS:
Time Frame: From initiation of study drug to 101 days of dosing discontinuation (assessed up to March 2017, approximately 16 months)
Description: The collection of nonserious AE information began at initiation of the study drug, and continued until Day 71. Monitoring of SAEs began from the date of the subject's written consent to participate in the study until Day 101. Nonserious AEs were followed to resolution or stabilization or reported as SAEs if they became serious. All SAEs that occurred with 101 days of dosing discontinuation were collected.
Groups:
- Belatacept Process E: Active Pharmaceutical Ingredient (API) of Belatacept manufactured by Process E
- Belatacept Process C: Active Pharmaceutical Ingredient (API) of Belatacept manufactured by Process C
Arm/Group | Belatacept Process E | Belatacept Process C
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/74 | 1/72
Other Adverse Events (participants affected / at risk) | 25/74 | 27/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Process E (N=74) | Belatacept Process C (N=72)
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept Process E (N=74) | Belatacept Process C (N=72)
Nausea (Gastrointestinal disorders) | 1 | 4
Nasopharyngitis (Infections and infestations) | 6 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 6
Headache (Nervous system disorders) | 11 | 21
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT02564497/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT02564497/SAP_001.pdf